CLINICAL TRIAL: NCT00577590
Title: Cyclotron Produced Isotopes in Biology and Medicine, Project 3: Specific Aim 1A and 1B Effects of Fatty Acid Delivery on Myocardial Metabolism and Function in Type 2 Diabetes (T2DM)
Brief Title: Effects of Fatty Acid Delivery on Heart Metabolism and Function in Type 2 Diabetes (T2DM
Acronym: T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 487
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type II
Keywords: Type II Diabetes Mellitus; Diabetes; PET; Heart Metabolism; Lovaza
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Metformin; Rosiglitazone; Omacor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metformin Alone (Placebo Comparator): Participants assigned to take Metformin alone.
  Interventions: Drug: Metformin
- Metformin and Rosiglitazone (Experimental): Participants assigned to take Metformin and Rosiglitazone
  Interventions: Drug: Metformin; Drug: Rosiglitazone
- Metformin and Lovaza (Experimental): Participants assigned to take Metformin and Lovaza
  Interventions: Drug: Metformin; Drug: Lovaza

INTERVENTIONS:
Drug: Metformin — Metformin is taken alone
  Other Names: Glumetza, Glucophage, Fortamet, Riomet
Drug: Rosiglitazone — Rosiglitizone is taken with Metformin
  Other Names: Advandia
  Arms: Metformin and Rosiglitazone
Drug: Lovaza — Lovaza is taken with Metformin
  Other Names: Omega-3 acid ethyl esters
  Arms: Metformin and Lovaza

SUMMARY:
Type 2 Diabetes Mellitus (T2DM) is a disease that interferes with the body's proper production and use of insulin, a hormone needed to convert sugar into usable energy. People with Type 2 Diabetes Mellitus (T2DM) are at a higher risk for certain cardiovascular diseases, including heart disease and stroke. Normal treatments for Type 2 Diabetes Mellitus (T2DM) target blood sugar levels only, but there is reason to believe that also targeting blood fat levels will improve both sugar metabolism and heart function in people with Type 2 Diabetes Mellitus, (T2DM.) This study will determine the effectiveness of blood-fat lowering treatments along with blood-sugar control treatments in improving heart function and symptoms of people with Type 2 Diabetes Mellitus(T2DM), and if this varies between men and women.

DETAILED DESCRIPTION:
Type 2 Diabetes Mellitus, (T2DM) is the most common type of diabetes. In Type 2 Diabetes Mellitus (T2DM), the body does not properly process sugars and, as a result, there is an excess amount of sugar in the blood. Eventually, the high blood sugar levels can lead to heart disease, nerve damage, kidney problems, or blindness. Typical Type 2 Diabetes Mellitus (T2DM) treatments target maintenance of blood sugar levels. Previous studies on Type 2 Diabetes Mellitus (T2DM) have indicated that in people who have high amounts of fats in the blood, the body relies more heavily on fats than sugars as an energy source. This dependence on fats for energy has been shown to have a negative effect on heart function. There is reason to believe that lowering the levels of fats in the blood will enhance the ability of the heart and the whole body to efficiently use both fats and sugars as energy sources. This study will evaluate the effectiveness of treatment strategies that are designed to reach target levels of sugar and fat in the blood for treating people with Type 2 Diabetes Mellitus (T2DM).

Participation in this double-blind study will last between 4 and 6 months. First, participants will undergo a medical screening and medication adjustment period, expected to last 6 months. The medical screening, lasting about 1 hour, will involve completing a medical history, physical exam, pregnancy test if applicable, and blood test to measure various factors that contribute to diabetes control. Participants will also be asked permission to store 1 tablespoon of their blood for up to 10 years to be used in future studies concerning genetics and heart energy metabolism. During the medication adjustment period, study physicians will adjust the participants' medications, offer advice on diabetes education and nutrition, and record any side effects from the medications. For newly diagnosed Type 2 Diabetes Mellitus (T2DM) participants, the study physician may recommend medication changes to assure a hemoglobin A1c (HgA1c) level of less than 7.5%. If participants have already achieved this level, they will be asked to continue present medications and to also begin taking the medication metformin for the 30 days before they undergo several imaging studies. Next, participants will complete routine tests that evaluate the pumping function of the heart, including an electrocardiogram (ECG) performed before and during exercise, a body composition study using a dual energy x-ray absorptiometry (DEXA) scan, and a magnetic resonance imaging (MRI) test. Each of these tests will last between 30 and 90 minutes.

After the qualifying tests, participants will return for the first of two separate imaging days that will include the same tests. The second imaging day will occur at the end of the medication period, approximately 2 months after the first imaging day. The first tests will be a whole body metabolism study and a heart metabolism imaging study, performed simultaneously. The whole body metabolism study will involve the injection of two tracers of metabolism, one for glucose and one for fatty acids. The heart metabolism imaging study will involve a positron-emission tomographic (PET) scan to take pictures of the heart and will include blood draws. The final imaging test will be a resting echocardiogram (ECHO) to measure heart function.

Following completion of the first day of imaging tests, participants will be randomly assigned to one of three possible treatment groups: Group A ,B, or C. Group A will take Metformin alone.Group B will take Metformin and Rosiglitazone. Group C will take Metformin and Lovaza. Participants will be seen monthly for the next 4 months, during which study medication will be distributed and blood pressure, heart rate, weight, and any side effects, such as lower extremity swelling, will be measured. If there is a noticeable increase in swelling, study physicians may adjust medication dosages. During visits at Months 2 and 4, blood samples will be taken to measure liver and organ function and HgA1c. At the completion of the 4-month medication treatment, participants will undergo repeat imaging tests. If needed, participants will be offered the opportunity to attend one or more follow-up visits to re-establish a medication routine.

ELIGIBILITY:
Inclusion Criteria:

* Meets Americans with Disabilities Act (ADA) criteria for T2DM; if newly diagnosed, must have fasting blood glucose greater than 126 mg/dl on two occasions, a random blood glucose greater than 200 mg/dl with symptoms, or a diagnostic oral glucose tolerance test
* Weight of less than 350 pounds
* Hemoglobin A1c of equal to or less than 7.5% at study entry or willing to go on one of the following therapies to achieve necessary percentage: metformin monotherapy greater than 1000 mg daily for at least 30 days or metformin greater than 1000 mg daily plus any combination of sulfonylurea, glipizide, or alpha-glucosidase inhibitor
* Blood pressure less than 140/90 mm Hg at study entry
* LDL level less than 130 mg/dL if on stable lipid lowering regimen
* Willing to undergo normal rest/stress (treadmill or dobutamine) echocardiogram
* If currently taking thyroid replacement therapy, must be on a stable dose of thyroid replacement and must have a thyroid function blood test that is in the normal range
* Willing to use an effective form of birth control throughout the study

Exclusion Criteria:

* Received therapy with an insulin sensitizer of the thiazolidinedione class within 6 months prior to study entry
* Required insulin therapy for more than 2 weeks in the year prior to study entry
* History of angina, heart attack, coronary artery bypass grafting (CABG), stroke, congestive heart failure (CHF), or peripheral vascular disease (PVD)
* Known coronary artery disease (CAD) with residual lesions of greater than 50%
* Current smoker
* Use or expected use of corticosteroids in any form
* Serum triglycerides greater than 400 mg/dl on a fasting sample at study entry
* Any contraindication to a thiazolidinedione (TZD) insulin sensitizer, metformin, or other drugs likely to be used during the study
* Liver disease with liver function test (LFT) greater than 2 times the upper limit of normal (ULN)
* Serum creatinine greater than 1.5 mg/dl for women and 1.6 mg/dl for men OR greater than 2+ proteinuria on urine dipstick

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2003-10; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gropler, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Harris MI, Flegal KM, Cowie CC, Eberhardt MS, Goldstein DE, Little RR, Wiedmeyer HM, Byrd-Holt DD. Prevalence of diabetes, impaired fasting glucose, and impaired glucose tolerance in U.S. adults. The Third National Health and Nutrition Examination Survey, 1988-1994. Diabetes Care. 1998 Apr;21(4):518-24. doi: 10.2337/diacare.21.4.518. PMID 9571335
- [Background] Grundy SM, Benjamin IJ, Burke GL, Chait A, Eckel RH, Howard BV, Mitch W, Smith SC Jr, Sowers JR. Diabetes and cardiovascular disease: a statement for healthcare professionals from the American Heart Association. Circulation. 1999 Sep 7;100(10):1134-46. doi: 10.1161/01.cir.100.10.1134. No abstract available. PMID 10477542
- [Background] Kannel WB, Hjortland M, Castelli WP. Role of diabetes in congestive heart failure: the Framingham study. Am J Cardiol. 1974 Jul;34(1):29-34. doi: 10.1016/0002-9149(74)90089-7. No abstract available. PMID 4835750
- [Background] Koskinen P, Manttari M, Manninen V, Huttunen JK, Heinonen OP, Frick MH. Coronary heart disease incidence in NIDDM patients in the Helsinki Heart Study. Diabetes Care. 1992 Jul;15(7):820-5. doi: 10.2337/diacare.15.7.820. PMID 1516498
- [Background] Abbott RD, Donahue RP, Kannel WB, Wilson PW. The impact of diabetes on survival following myocardial infarction in men vs women. The Framingham Study. JAMA. 1988 Dec 16;260(23):3456-60. PMID 2974889
- [Derived] Peterson LR, Saeed IM, McGill JB, Herrero P, Schechtman KB, Gunawardena R, Recklein CL, Coggan AR, DeMoss AJ, Dence CS, Gropler RJ. Sex and type 2 diabetes: obesity-independent effects on left ventricular substrate metabolism and relaxation in humans. Obesity (Silver Spring). 2012 Apr;20(4):802-10. doi: 10.1038/oby.2011.208. Epub 2011 Aug 4. PMID 21818149

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin and Lovaza: Participants assigned to take metformin and Lovaza
  Lovaza: Dosage of 4 g to be taken daily for 2 months
  Metformin: Dosage of at least 1000 mg to be taken daily for 4 months
- Metformin: Participants assigned to take metformin and placebo
  Metformin: Dosage of at least 1000 mg to be taken daily for 4 months
- Metformin and Rosiglitazone: Patients received Metformin and Rosiglitizone
Period: Overall Study
Arm/Group | Metformin and Lovaza | Metformin | Metformin and Rosiglitazone
Started | 28 | 27 | 23
Completed | 28 | 27 | 23
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Metformin and Rosiglitizone: Participants assigned to take Metformin and Rosiglitizone
- Total: Total of all reporting groups
Arm/Group | Metformin and Lovaza | Metformin | Metformin and Rosiglitizone | Total
Number analyzed (Participants) | 28 | 27 | 23 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 27 | 23 | 78
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 15 | 43
  Male | 15 | 12 | 8 | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 27 | 23 | 78

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Plasma Triglycerides
Time Frame: Baseline and 3 months
Population: Data presented are stratified by sex
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Metformin and Lovaza | Metformin | Metformin and Rosiglitazone
Number analyzed (Participants) | 28 | 27 | 23
percent change
  Plasma triglycerides women: number analyzed (Participants) | 13 | 15 | 15
  Plasma triglycerides women | -2.0 (12) | 16.0 (30) | -5.0 (15)
  Plasma triglycerides men: number analyzed (Participants) | 15 | 12 | 8
  Plasma triglycerides men | -5.0 (12) | -10.0 (5) | 1.0 (12)

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Metformin and Lovaza | Metformin | Metformin and Rosiglitizone
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 0/23
Other Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 0/23

LIMITATIONS AND CAVEATS:
There were no limitations or caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes